CLINICAL TRIAL: NCT04270643
Title: Trial of High-Dose Vitamin D in the Treatment of Complicated Severe Acute Malnutrition
Acronym: ViDiSAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University of the Punjab (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ViDiSAM
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): Two oral doses of 5 mg (200,000 international units) vitamin D3 in 1 ml ethyl oleate, given at baseline and two weeks thereafter
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Two oral doses of 1 ml ethyl oleate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — ATC code A11CC05 (cholecalciferol)
  Arms: Vitamin D
Dietary Supplement: Placebo — Ethyl oleate
  Arms: Placebo

SUMMARY:
This double-blind randomized placebo-controlled controlled trial will test the hypothesis that administration of high-dose oral vitamin D supplementation to children in Lahore, Pakistan, who are recovering from complicated severe acute malnutrition will safely accelerate weight gain (primary outcome) and enhance neurodevelopment, muscle mass accumulation, resolution of systemic inflammation and antimicrobial immune function (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Consent of parent / guardian
* Age 6-59 months at enrolment
* Diagnosis of complicated SAM at the point of hospital admission as defined by the World Health Organisation.
* Medical team managing the child has made the decision to discharge the child from inpatient care

Exclusion Criteria:

* Ingestion of a dose of vitamin D>200,000 IU (5 mg) in the last 3 months
* Known diagnosis of primary hyperparathyroidism or sarcoidosis (i.e. conditions pre-disposing to vitamin D hypersensitivity)
* Known neurodevelopmental disorder (e.g. cerebral palsy)
* HIV infection
* Taking anti-tuberculosis treatment
* Inability to assess child's developmental status at baseline using the Malawi Development Assessment Tool
* Signs of rickets
* Corrected serum calcium concentration >2.65 mmol/L on blood sample taken during the current hospital admission

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 259 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Mean weight-for-height/length z-score | 2 months

SECONDARY OUTCOMES:
Mean weight-for-height/length z-score | 6 months
Mean weight-for-age z-score | 2 and 6 months
Mean height/length-for-age z-score | 2 and 6 months
Mean head circumference-for-age z-score | 2 and 6 months
Mean mid-upper arm circumference | 2 and 6 months
Mean change in overall and domain-specific (gross motor, fine motor, language and social) neurodevelopmental scores, Malawi Developmental Assessment Tool | 2 and 6 months
Mean fat mass index | 2 and 6 months
Mean fat-free mass index | 2 and 6 months
Proportion of participants experiencing relapse of severe acute malnutrition | 6 months
Proportion of participants readmitted to hospital due to any cause | 6 months
Antimicrobial immune function (concentrations of inflammatory mediators in supernatants of whole blood stimulated with lipo-polysaccharide, zymosan and heat-killed Salmonella typhi) | 2 and 6 months
Serum concentrations of albumin, C-reactive protein, 25-hydroxyvitamin D, total alkaline phosphatase, parathyroid hormone, ferritin and hepcidin | 2 and 6 months
Mean haemoglobin concentration, full blood count | 2 and 6 months
Mean corpuscular volume, full blood count | 2 and 6 months
Mean corpuscular haemoglobin concentration, full blood count | 2 and 6 months
Mean neutrophil count, full blood count | 2 and 6 months
Mean lymphocyte count, full blood count | 2 and 6 months
Mean monocyte count, full blood count | 2 and 6 months
Faecal concentrations of inflammatory markers (myeloperoxidase, neopterin and alpha-1 antitrypsin) | 2 and 6 months
Faecal microbiome composition | 2 and 6 months
Proportion of participants dying | 6 months
Incidence of serious adverse events | 6 months
Incidence of adverse reactions | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Sir Ganga Ram Hospital, Lahore
  - THQ Hospital, Lahore

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with other researchers subject to terms of Data Transfer Agreement and IRB approval
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 2 years after completion of the trial

REFERENCES:
- [Derived] Saleem J, Zakar R, Butt MS, Kaleem R, Chaudhary A, Chandna J, Jolliffe DA, Piper J, Abbas Z, Tang JCY, Fraser WD, Freemantle N, Prendergast AJ, Martineau AR. High-dose vitamin D3 to improve outcomes in the convalescent phase of complicated severe acute malnutrition in Pakistan: a double-blind randomised controlled trial (ViDiSAM). Nat Commun. 2025 Mar 15;16(1):2554. doi: 10.1038/s41467-025-57803-9. PMID 40089464